CLINICAL TRIAL: NCT07047469
Title: Ultrasound-assisted Spinal Anesthesia in Midline Versus Paramedian Approach in Adult Orthopedic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Areej Mohamed Abdelkader, Resident, Department of Anesthesia, Intensive Care and Pain management, Faculty of Medicine, Sohag University, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Soh-Med--25-6-16MS
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Anesthesia; Functional
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (1): spinal anesthesia with median approach (Active Comparator): patients undergoing orthopedic surgery will receive spinal anesthesia with median approach under ultrasound guided techniques
  Interventions: Procedure: Group (1): spinal anesthesia with median approach
- Group (2): spinal anesthesia with paramedian approach (Active Comparator): patients undergoing orthopedic surgery will receive spinal anesthesia with paramedian approach under ultrasound guided techniques
  Interventions: Procedure: Group (2): spinal anesthesia with paramedian approach

INTERVENTIONS:
Procedure: Group (1): spinal anesthesia with median approach — patients undergoing orthopedic surgery will receive spinal anesthesia with median approach under ultrasound guided techniques
  Arms: Group (1): spinal anesthesia with median approach
Procedure: Group (2): spinal anesthesia with paramedian approach — patients undergoing orthopedic surgery will receive spinal anesthesia with paramedian approach under ultrasound guided techniques
  Arms: Group (2): spinal anesthesia with paramedian approach

SUMMARY:
This study aims to compare between the two methods (midline and paramedian approach of spinal anesthesia guided by ultrasound) by the number of needle passes required to successful dural puncture.

ELIGIBILITY:
Inclusion Criteria:

* Patients will perform orthopedic surgery
* Physical state I or II according to ASA classification
* Age between (18 - 50 )
* Body mass index less than 30

Exclusion Criteria:

* Patient refusal .
* Local infection at the puncture site .
* Allergy to any of the drugs to be administrated .
* Old age patients
* Obese patients
* Previous spinal surgery .
* Spinal stenosis .
* Multiple sclerosis .
* Coagulopathy.
* Hypovolemia .
* Systemic infection .
* Aortic stenosis .
* Spina bifida and back deformity .

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
The severity of back pain in patients that will receive spinal anesthesia by median versus paramedian approach | 24 hours, 72 hours, and 1 week after spinal anesthesia.
  pain measurement by numerical rating scale (NRS)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Zeng W, Shi Y, Zheng Q, Du S. Ultrasound-assisted modified paramedian technique for spinal anesthesia in elderly. BMC Anesthesiol. 2022 Jul 30;22(1):242. doi: 10.1186/s12871-022-01751-0. PMID 35907825
- [Background] Singh B, Sohal AS, Singh I, Goyal S, Kaur P, Attri JP. Incidence of Postspinal Headache and Low Backache Following the Median and Paramedian Approaches in Spinal Anesthesia. Anesth Essays Res. 2018 Jan-Mar;12(1):186-189. doi: 10.4103/aer.AER_139_17. PMID 29628579
- [Background] Wilson JM, Farley KX, Erens GA, Guild GN 3rd. General vs Spinal Anesthesia for Revision Total Knee Arthroplasty: Do Complication Rates Differ? J Arthroplasty. 2019 Jul;34(7):1417-1422. doi: 10.1016/j.arth.2019.03.048. Epub 2019 Mar 28. PMID 31005435